CLINICAL TRIAL: NCT00146731
Title: Treating Malaria During Pregnancy: A Randomized Trial of Potential Options for Treatment in an Area of High Drug Resistance in Tanzania
Brief Title: A Trial of Antimalarial Drugs Used in Pregnancy in Tanzania
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITCRVG04
Record Dates: First submitted 2005-09-05; First posted 2005-09-07 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
Keywords: malaria; pregnancy; treatment; Africa; Tanzania
MeSH Terms: conditions — Malaria | interventions — Amodiaquine; Artesunate; chloroguanil, dapsone drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: SP
Drug: SP + amodiaquine
Drug: AQ + artesunate
Drug: chlorproguanil-dapsone

SUMMARY:
Pregnant women are vulnerable to malaria, with significant implications both for their health and for the pregnancy. Sulfadoxine-pyrimethamine (SP) is currently the first line drug for the treatment of malaria in pregnancy in Tanzania and surrounding countries, but resistance is emerging rapidly. Alternative drugs must be found, and new drugs and drug combinations are being recommended by many for deployment as first line treatment at the point that SP resistance forces a policy change. However, there are few data on the safety and efficacy of these combinations in pregnant women. This randomised trial aims to assess efficacy and safety, including birth outcome, in pregnant women with malaria in the second or third trimesters. A total of 900 pregnant women will be randomised either to standard treatment (SP) or to one of three potential drugs, or drug combinations recently recommended by a WHO expert panel. These will be SP-amodiaquine, chlorproguanil-dapsone (Lapdap), and amodiaquine-artesunate. Primary outcome will be treatment failure. Secondary outcomes will include 28 day slide clearance, maternal side effects, foetal viability and birth outcome.

DETAILED DESCRIPTION:
The objectives of this study are to assess the therapeutic efficacy and safety of SP as the current first line drug, and three other potential alternative combinations in treating uncomplicated falciparum malaria during pregnancy, in an area with appreciable levels of SP resistance and rising HIV seroprevalence. Specifically the study will compare the clinical and parasitological response to and the side effects of the following drug regimes:

1. SP
2. SP + amodiaquine (SPAQ)
3. Chlorproguanil+dapsone (Lapdap)
4. Amodiaquine + artesunate (AQAS)

TRIAL DESIGN

Primary end point

The primary end-point of the trial will be treatment failure. This will be defined as:-

Any of:

1. a need for rescue treatment due to clinical deterioration defined by altered sensorium, convulsions, persistent vomiting, renal impairment, respiratory distress, a fall in Hb below 75g/dl, or in cases where initial haemoglobin was less than 9 g/dl a drop of 20% from the starting Hb if the initial Hb was less than 9g/dl, at any time during admission;
2. persistence of fever with parasitaemia on day 32;
3. increasing parasite load on day 3;
4. failure to clear parasites on day 7;
5. rescue medication for recurrent malaria before day 14;
6. slide parasite positivity at day 14.

Secondary endpoints

Secondary endpoints will include the following:-

1. Incidence of foetal death during treatment, defined as absence of foetal heartbeat assessed by Doppler
2. Hypoglycaemia requiring treatment
3. Parasite recrudescence or re-infection on day 28
4. Parasite clearance on day 3
5. Level of recovery of haemoglobin on day 14
6. Fever clearance time
7. Incidence of perinatal and neonatal mortality, assessed 4-6 weeks after due date of delivery
8. Clinically apparent neonatal abnormality, assessed 4-6 weeks after due date of delivery
9. Placental malaria
10. Preterm delivery
11. Other adverse events during treatment

The trial

1. This will be a randomized controlled trial with four arms
2. The slide reader assessing the primary endpoint will be blind to treatment allocation, and analysis will be performed by intention-to-treat
3. Direct Observed Therapy (DOT) of all doses of study regimens will be employed
4. Drug doses packed in blister packs, labelled with the patient number will be used where possible.
5. Selection and Withdrawal of Patients

Pregnant women with mild-moderate, slide proven, falciparum malaria will be recruited from the Antenatal wing (ANC) of the Maternal and Child Health (MCH) clinic at Muheza (Teule) Hospital. Pregnant women from Muheza Township and surrounding villages attend this clinic. Nurses attending the clinic will interview all febrile women and women with a recent (past 24 hours) history of fever and those with a probable diagnosis of malaria will be referred to the study team. Those with signs/symptoms of mild-moderate anaemia will also be referred. All referrals will be re-interviewed and examined by the Medical Officer of the study team to exclude concomitant infection(s). Duplicate thick and thin blood smears will be made, Giemsa stained at pH 7.2, and examined microscopically. The consent form will be administered to those meeting the inclusion criteria and they will be enrolled upon consenting.

Inclusion criteria

A pregnant woman who has:-

either a positive blood smear for P.falciparum with at least 1000 asexual parasites/uL in an asymptomatic woman or any of the following symptoms within 2 days prior to consultation: history of fever; headache, vomiting, chills/rigors, and/or any of the following signs: temperature >37.50C and <39.50C, Hb >5 and <9 g/dl) together with P.falciparum parasitaemia at any density

and (in both cases) the following:

1. has no exclusion criterion (see below)
2. is 14-34 weeks pregnant on the day of attending the ANC clinic or OPD;
3. has a viable foetus, defined by presence of foetal heartbeat by sonicaid or pinnard (foetal heartbeat is not heard until 14 weeks)
4. is able to take study drugs by the oral route
5. is able to attend stipulated days for follow up clinic and provide specimens
6. gives informed written or witnessed verbal consent to participate by herself, and also through her parent/guardian if aged <15 years (in conformity to Tanzania Law)

Those > 34 weeks are excluded because they are close to term and may deliver during the 28 day follow up period.

Exclusion criteria

Exclusion criteria include:-

1. severe and complicated forms of malaria (as defined by WHO, 1996);
2. pregnancy in the first trimester;
3. a mixed plasmodial infection;
4. complicated pregnancy e.g. signs/symptoms of toxaemia of pregnancy;
5. 23 or more abortions or stillbirths;
6. presence of concomitant disease masking assessment of the response to treatment ;
7. an intake of drugs contraindicated in pregnancy e.g. tetracycline, cotrimoxazole or a macrolide antibiotic;
8. an intake of drugs with effective antimalarial activity within the last 2 weeks.
9. significantly abnormal baseline haematology (except anaemia) or clinical chemistry parameters e.g. laboratory evidence of renal impairment (serum creatinine >2 mg/dl) or of hepatitis (alanine aminotransferase ALT>5 times upper limit of normal);
10. previous participation in the study: Women having a second episode of malaria after completing the 28-day follow up will have details recorded and offered quinine but not be re-enrolled.
11. multiple gestation pregnancies eg twins
12. Mother aged 38 years or above

Patients with malaria who do not enter the trial because they fulfil an exclusion criterion will be treated in the optimum way decided by the attending physician. In general, those with severe disease will receive parenteral quinine whilst those with mild disease will receive SP.

Withdrawal criteria

Withdrawal criteria will include:-

1. withdrawal of consent or non-compliance with assigned study regimen;
2. appearance of other species of Plasmodium;
3. vomiting within one hour after re-dosing;
4. protocol violation.

   If it is necessary to withdraw a patient during the treatment phase, administration of the study drug will be discontinued. If the patient is still parasitaemic, quinine will be given as a rescue therapy unless there are clinical reasons to use another drug. For withdrawals outside the treatment phase the team will carry out all the safety and efficacy assessment measurements that would have been carried out at the next scheduled visit and the same will apply at delivery (unless the patient is lost to follow up).
5. Patients who fail on treatment will be treated with rescue treatment and counted as treatment failures (see above).

TREATMENT OF PATIENTS

Study regimens

Study drugs will be purchased or sourced from reputable sources with Good Manufacturing Practice (GMP). Dosages will be based on the body weight (kg) of the patient and the schedule will be as below.

1. SP (sulfadoxine 25mg/kg stat)(SP)
2. SP (sulfadoxine 25mg/kg stat) + Amodiaquine (10mg/kg x 3 days) (SPAQ)
3. Chlorproguanil-dapsone (1.2 mg/kg and 2.4 mg/kg respectively 3 days) [Lapdap]
4. Amodiaquine (10mg/kg x 3 days) + Artesunate (4mg/kg x 3 days) (AQAS)

ELIGIBILITY:
Inclusion Criteria:

A pregnant woman who has either a positive blood smear for P.falciparum with at least 1000 asexual parasites/uL in an asymptomatic woman

or any of the following symptoms within 2 days prior to consultation:

* history of fever;
* headache,
* vomiting,
* chills/rigors,
* and/or any of the following signs: temperature >37.50C and <39.50C, Hb>5 and <9 g/dl together with P.falciparum parasitaemia at any density

and (in both cases) the following:

1. Has no exclusion criterion (see below);
2. Is 14-34 weeks pregnant on the day of attending the ANC clinic or OPD;
3. Has a viable foetus, defined by presence of foetal heartbeat by sonicaid or pinnard (foetal heartbeat is not heard until 14 weeks);
4. Is able to take study drugs by the oral route;
5. Is able to attend stipulated days for follow up clinic and provide specimens;
6. Gives informed written or witnessed verbal consent to participate by herself, and also through her parent/guardian if aged <15 years (in conformity to Tanzania Law).

Exclusion Criteria:

1. Severe and complicated forms of malaria (as defined by WHO, 1996);
2. Pregnancy in the first trimester;
3. A mixed plasmodial infection;
4. Complicated pregnancy, e.g. signs/symptoms of toxaemia of pregnancy;
5. 23 or more abortions or stillbirths;
6. Presence of concomitant disease masking assessment of the response to treatment ;
7. An intake of drugs contraindicated in pregnancy, e.g. tetracycline, cotrimoxazole or a macrolide antibiotic;
8. An intake of drugs with effective antimalarial activity within the last 2 weeks.
9. Significantly abnormal baseline haematology (except anaemia) or clinical chemistry parameters, e.g. laboratory evidence of renal impairment (serum creatinine >2 mg/dl) or of hepatitis (alanine aminotransferase [ALT] >5 times upper limit of normal);
10. Previous participation in the study: Women having a second episode of malaria after completing the 28-day follow up will have details recorded and offered quinine but not be re-enrolled.
11. Multiple gestation pregnancies, eg twins
12. Mother aged 38 years or above

Ages: 15 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 310 (Actual)
Dates: Start 2004-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary end-point of the trial will be treatment failure. This is defined above.

SECONDARY OUTCOMES:
Incidence of foetal death during treatment, defined as absence of foetal heartbeat assessed by Doppler
Hypoglycaemia requiring treatment
Parasite recrudescence or re-infection on day 28
Parasite clearance on day 3
Level of recovery of haemoglobin on day 14
Fever clearance time
Incidence of perinatal and neonatal mortality, assessed 4-6 weeks after due date of delivery
Clinically apparent neonatal abnormality, assessed 4-6 weeks after due date of delivery
Placental malaria
Preterm delivery
Other adverse events during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Theonest K Mutabingwa, MD PhD, Study Director — LSHTM/NIMR; Christopher JM Whitty, FRCP, Principal Investigator — London School of Hygiene and Tropical Medicine; Daniel Chandramohan, MD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Muheza Designated District Hospital, Muheza, Tanga, Tanzania

REFERENCES:
- [Derived] Mutabingwa TK, Muze K, Ord R, Briceno M, Greenwood BM, Drakeley C, Whitty CJ. Randomized trial of artesunate+amodiaquine, sulfadoxine-pyrimethamine+amodiaquine, chlorproguanal-dapsone and SP for malaria in pregnancy in Tanzania. PLoS One. 2009;4(4):e5138. doi: 10.1371/journal.pone.0005138. Epub 2009 Apr 8. PMID 19352498